CLINICAL TRIAL: NCT04251897
Title: Novel Support Surface Based on Smart Materials to Alleviate Pressure Ulcer Formation During the Rehabilitation of Immobile Patients
Brief Title: Novel Support Surface to Alleviate Pressure Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: DSRB 2019/00002
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Immobility Syndrome; Pressure Ulcer; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care mattress (Active Comparator): Patient will have 2 days to familiarize with the novel support surface. Patient will be on standard care mattress. They will be turned over every 2 hours for 3 days.
  Interventions: Device: Novel support surface
- Novel support surface (Experimental): After the standard care mattress, the same patient will be placed on novel support surface. They will be turned over every 2 hours for 3 days.
  Patient will then continue with the novel support surface and turned every 3 hours for 3 days.
  They will then continue with the novel support surface and turned every 4 hours for 3 days.
  Interventions: Device: Novel support surface

INTERVENTIONS:
Device: Novel support surface — This is a magnetorheological elastomer that can dynamically redistribute the pressure over a bony prominence to be lower than the critical closing pressure while at the same time providing sufficient support.

SUMMARY:
A prototype support surface has been designed which aims to successfully redistributes the pressures exerted and provides sufficient support to human soft tissue

We want to prove the effectiveness of the prototype support surface by enlisting patients in a clinical trial, where we will assess the presence of pressure ulcers, and the ability of the patients to tolerate the support surface, and also measure the pressure over time and compare them to when the patients are using standard mattresses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be immobile as assessed on the braden scale.
2. Patients must require 2 hourly turning
3. Age 21-85

Exclusion Criteria:

1. No existing pressure ulcers
2. No active infections, fever, or medical conditions that require constant medical attention.
3. They must also not have severe incontinence requiring the change of diapers more frequently than 4 hours
4. No significant cognitive impairment
5. Pregnant women will be excluded from the study

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
PTAUC | For a maximum of 14 days (duration of trial)
  pressure-time area under curve
Pressure sores - NPUAP (National Pressure Ulcer Advisory Panel) grade | For a maximum of 14 days (duration of trial)
  If pressure sores are present, they will be graded based on the NPUAP grade from 1-4. Location will also be recorded.

SECONDARY OUTCOMES:
Patient's comfort | For a maximum of 14 days (duration of trial)
  Patient comfort measured on a visual analogue scale (1- 10)
Discomfort or pain | For a maximum of 14 days (duration of trial)
  Presence of discomfort or pain at high risk pressure points. This will be asked of patients, and will be scored as yes or no.
Suggestions | For a maximum of 14 days (duration of trial)
  This will be a qualitative open-ended question for patient's verbatim report or suggestions

CONTACTS AND LOCATIONS:
Overall Officials: Chin Jung Wong, MD, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital Rehabilitation Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No